CLINICAL TRIAL: NCT01174875
Title: Developmental Pathways to Health and Disease: Metabolic, Neurodevelopmental and Related Outcomes
Brief Title: Growing Up in Singapore Towards Healthy Outcomes
Acronym: GUSTO
Status: Active, not recruiting | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: KK Women's and Children's Hospital (Other Government); Institute for Human Development and Potential (IHDP), Singapore (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, Obstetrics & Gynaecology, Professor Chong Yap Seng, National University Hospital, Singapore
Other Study IDs: CIRB 2019/2655/E; NMRC/TCR/004-NUS/2008 (Other Grant/Funding Number: National Medical Research Council); NMRC/TCR/012-NUHS/2014 (Other Grant/Funding Number: National Medical Research Council); MOH-000504 (Other Grant/Funding Number: National Medical Research Council)
Record Dates: First submitted 2010-07-01; First posted 2010-08-04 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Diseases; Neurological and Mental Health Conditions; Genetic Predisposition; Skin Condition; Environmental Exposure; Socioeconomic Factors; Psychology, Social
Keywords: Epigenetics; Development; Metabolic; Neurodevelopment; Cohort Study; Birth Cohort; Longitudinal Study; Pregnancy; Growth; Developmental Origins of Health and Disease; DOHaD; Epidemiology; Maternal Health; Infant Health; Child Health; Health Outcomes; Postnatal Exposure; Perinatal Exposure; Environmental Factors; Nutrition; Genetics
MeSH Terms: conditions — Metabolic Diseases; Neurologic Manifestations; Genetic Predisposition to Disease; Skin Diseases; Developmental Origins of Health and Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of human biological materials such as blood, cord, cord blood, placenta, vaginal swabs, rectal swabs, skin (vulva and breast) swabs, nasal swab, skin microbiome samples, breast milk, hair, saliva, buccal swabs, exfoliated milk teeth, urine, stool, dental plaque/biofilm and skin samplings (using ceramic discs, skin tapes and swabs),
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant mothers, infants and children: Women in their early pregnancy who are attending the first trimester antenatal ultrasound scan at the public maternity units at KK Women's and Children's Hospital (KKH) and National University Hospital (NUH). Only women age 18 years and above who are Singapore Citizens or Singapore Permanent Residents. Participants have to intend to eventually deliver in NUH or KKH and to reside in Singapore for the next 5 years. Willingness to donate cord, cord blood and placenta. The fetus should be racially homogenous with both sets of grandparents of the same ethnicity. Babies born from these mothers will be followed up until the child is at least 20 years of age.

SUMMARY:
This study aims to examine the role of genetic and epigenetic factors, maternal nutrition, lifestyle, emotional health, and other environmental factors in pregnancy or postpartum period that can influence future maternal risk of metabolic and mental wellness, including body weight changes. The study will recruit women in early pregnancy and later follow their children after birth, tracking both the mother and child until the child reaches at least 20 years of age.

DETAILED DESCRIPTION:
The dramatic emergence of non-communicable diseases (NCDs) in Asia has coincided with the rapid socioeconomic and nutritional transition taking place in the region, with the prevalence of diabetes rising five-fold in Singapore in less than four decades. One unique aspect of the epidemic has been the significant ethnic differences in predisposition to diabetes among Asians and in the ethnic variation between BMI and the risk of developing insulin resistance, a precursor to type 2 diabetes. Apart from genetic factors, dietary, lifestyle and cultural factors might have influenced the developmental programming through effects on the mechanisms associated with developmental plasticity. A center piece of this study is to examine how epigenetic changes at birth both reflects past developmental influences and, in association with other factors, influences future trajectories of development and its relationship to NCDs. Also factors active during childhood - especially the first 1000 days of life - will be focused upon. The longitudinal GUSTO birth cohort study allows us to examine associations among genetic, environmental and lifestyle interactions in the three distinct ethnic groups, Chinese, Malays and Indians, present in the Singaporean population. Participants have been followed up for their pregnancy outcome, fetal growth and offspring development. In continuation of this research, participants will continue to be followed up through their adolescence phase from the age of 10 to 20 years.

Data will be collected through questionnaires and measurements.

* Questionnaires may be related to socioeconomic factors, healthcare expenses, diet, medical history, behaviour, cognition, lifestyle, sleep, health status, social-emotion factors, and home environment.
* Body measurements such as height, weight, blood pressure, body composition analysis involving bioelectrical impedance analysis (BIA), grip strength.
* Dental examination
* Child pubertal assessments
* Skin clinical assessment and digital photography for assessment of acne presence and severity
* Monitoring physical activity level and sedentary behaviour by using an accelerometer
* Using mobile phone app to collect information about your child's mobile phone usage patterns, activities etc.
* Collection of samples e.g. blood, buccal swabs, saliva, hair, urine, stool, skin samples, oral specimen such as exfoliated milk teeth, dental plaque and tongue biofilms

ELIGIBILITY:
Inclusion Criteria of Mother Participants:

* Women 18 years and above
* Pregnant women attending the first visit (< 14 weeks GA) at the maternity units of KKH and NUH
* Singapore citizens or Singapore Permanent Residents
* Currently resident in mainland Singapore
* Intention to eventually deliver in KKH or NUH
* Intention to reside in Singapore for the next 5 years
* Intention to donate cord, cord blood and placenta
* The fetus should be racially homogenous with both sets of grandparents of the same ethnicity

Exclusion Criteria of Mother Participants:

* Women whose pregnancies end in miscarriages will be excluded
* Pregnant women on chemotherapy
* Exclude women with significant medical conditions e.g. Type 1 diabetes mellitus, psychosis etc.
* Exclude women on certain medications - e.g. psychotropic drugs.
* Mixed marriages will be excluded

Babies born from these mothers will be invited to participate and followed up until the child is at least 20 years of age.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women attending their first-trimester antenatal visit at public maternity units in KKH and NUH, along with their children born from the indexed pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 1247 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Roles of fetal, developmental and epigenetic factors in pathways to disease | Perinatal
  To evaluate the role of fixed genetic risk variants, modifiable epigenetic markers, circulating metabolites and hormones in blood, and host-microbe interactions which can reflect past developmental influences, and in association with other factors, affect future trajectories of development and its relationship to NCDs.

SECONDARY OUTCOMES:
Influence of prenatal and early postnatal factors on child health | During pregnancy and infancy period
  To examine the role of maternal nutrition, lifestyle, emotional health, and other environmental factors in infancy that can influence the development of phenotypes in childhood which confer risk for later metabolic and mental disorders.
Effect of factors in pregnancy and early postpartum period on maternal health | During pregnancy and postpartum period
  To examine the role of maternal nutrition, lifestyle, emotional health, and other environmental factors in pregnancy or postpartum period that can influence future maternal risk of metabolic disorders, including body weight changes.
Influence genetic and epigenetics factors in combination with lifestyle on child health | Childhood and Adolescence up to age 20
  To examine the role of genetic and epigenetic factors, lifestyle (physical activity and dietary intake), growth trajectories and other environmental factors that can influence the development of phenotypes in childhood which confer risk for later metabolic and mental disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Yap Seng Chong, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soh SE, Tint MT, Gluckman PD, Godfrey KM, Rifkin-Graboi A, Chan YH, Stunkel W, Holbrook JD, Kwek K, Chong YS, Saw SM; GUSTO Study Group. Cohort profile: Growing Up in Singapore Towards healthy Outcomes (GUSTO) birth cohort study. Int J Epidemiol. 2014 Oct;43(5):1401-9. doi: 10.1093/ije/dyt125. Epub 2013 Aug 2. No abstract available. PMID 23912809
- [Derived] Pang WW, Geddes DT, Lai CT, Michael N, Huang J, Chan YH, Cheong CY, Fok D, Pundir S, Ng S, Vickers MH, Chua MC, Tan KH, Godfrey KM, Shek LP, Chong YS, Eriksson JG, Chan SY, Wlodek ME. The prospective associations of fetal growth-related pregnancy complications with subsequent breastfeeding duration and markers of human milk production. Am J Clin Nutr. 2025 Feb;121(2):478-487. doi: 10.1016/j.ajcnut.2024.11.008. Epub 2024 Nov 13. PMID 39542219
- [Derived] Han MX, Nadarajan R, Wang N, Kee MZL, Lim S, Sagar YK, Chow B, Tan AP, Cheon BK, Ang YS, Zhou JH, Chen HY, Chong YS, Gluckman PD, Meaney MJ, Law EC. Maternal Depressive Symptoms and Risk for Childhood Depression: Role of Executive Functions. J Am Acad Child Adolesc Psychiatry. 2025 Aug;64(8):946-958. doi: 10.1016/j.jaac.2024.08.503. Epub 2024 Oct 16. PMID 39419473
- [Derived] Padmapriya N, Bernard JY, Tan SYX, Chu AHY, Goh CMJL, Tan SL, Shek LP, Chong YS, Tan KH, Chan SY, Yap F, Godfrey KM, Lee YS, Meaney MJ, Eriksson JG, Tan CS, Law EC, Muller-Riemenschneider F. The prospective associations of 24-hour movement behaviors and domain-specific activities with executive function and academic achievement among school-aged children in Singapore. Front Public Health. 2024 Sep 4;12:1412634. doi: 10.3389/fpubh.2024.1412634. eCollection 2024. PMID 39296832
- [Derived] Xu J, Duar RM, Quah B, Gong M, Tin F, Chan P, Sim CK, Tan KH, Chong YS, Gluckman PD, Frese SA, Kyle D, Karnani N. Delayed colonization of Bifidobacterium spp. and low prevalence of B. infantis among infants of Asian ancestry born in Singapore: insights from the GUSTO cohort study. Front Pediatr. 2024 Jun 10;12:1421051. doi: 10.3389/fped.2024.1421051. eCollection 2024. PMID 38915873
- [Derived] Padmapriya N, Fogel A, Tan SYX, Goh CMJL, Tan SL, Chia A, Chu AHY, Chong YS, Tan KH, Chan SY, Yap F, Godfrey KM, Lee YS, Eriksson JG, Tan CS, Bernard JY, Muller-Riemenschneider F. The cross-sectional and prospective associations of parental practices and environmental factors with 24-hour movement behaviours among school-aged Asian children. Int J Behav Nutr Phys Act. 2024 Mar 4;21(1):27. doi: 10.1186/s12966-024-01574-x. PMID 38438945
- [Derived] Chia A, Toh JY, Natarajan P, Cai S, Ong YY, Descarpentrie A, Lioret S, Bernard JY, Muller-Riemenschneider F, Godfrey KM, Tan KH, Chong YS, Eriksson JG, Chong MF. Trajectories of lifestyle patterns from 2 to 8 years of age and cardiometabolic risk in children: the GUSTO study. Int J Behav Nutr Phys Act. 2024 Jan 26;21(1):9. doi: 10.1186/s12966-024-01564-z. PMID 38279175
- [Derived] Ong YY, Pang WW, Michael N, Aris IM, Sadananthan SA, Tint MT, Liang Choo JT, Ling LH, Karnani N, Velan SS, Fortier MV, Tan KH, Gluckman PD, Yap F, Chong YS, Godfrey KM, Chan SY, Eriksson JG, Chong MF, Wlodek ME, Lee YS. Timing of introduction of complementary foods, breastfeeding, and child cardiometabolic risk: a prospective multiethnic Asian cohort study. Am J Clin Nutr. 2023 Jan;117(1):83-92. doi: 10.1016/j.ajcnut.2022.10.021. Epub 2022 Dec 21. PMID 36789947
- [Derived] Mir SA, Chen L, Burugupalli S, Burla B, Ji S, Smith AAT, Narasimhan K, Ramasamy A, Tan KM, Huynh K, Giles C, Mei D, Wong G, Yap F, Tan KH, Collier F, Saffery R, Vuillermin P, Bendt AK, Burgner D, Ponsonby AL, Lee YS, Chong YS, Gluckman PD, Eriksson JG, Meikle PJ, Wenk MR, Karnani N. Population-based plasma lipidomics reveals developmental changes in metabolism and signatures of obesity risk: a mother-offspring cohort study. BMC Med. 2022 Jul 25;20(1):242. doi: 10.1186/s12916-022-02432-y. PMID 35871677
- [Derived] Kumar M, Ang LT, Ho C, Soh SE, Tan KH, Chan JKY, Godfrey KM, Chan SY, Chong YS, Eriksson JG, Feng M, Karnani N. Machine Learning-Derived Prenatal Predictive Risk Model to Guide Intervention and Prevent the Progression of Gestational Diabetes Mellitus to Type 2 Diabetes: Prediction Model Development Study. JMIR Diabetes. 2022 Jul 5;7(3):e32366. doi: 10.2196/32366. PMID 35788016
- [Derived] Loo EXL, Ooi DSQ, Ong M, Ta LDH, Lau HX, Tay MJY, Yap QV, Chan YH, Tham EH, Goh AEN, Van Bever H, Teoh OH, Eriksson JG, Chong YS, Gluckman P, Yap FKP, Karnani N, Xu J, Tan KML, Tan KH, Lee BW, Kramer M, Shek LP, Meaney MJ, Broekman BFP. Associations Between Eczema and Attention Deficit Hyperactivity Disorder Symptoms in Children. Front Pediatr. 2022 Mar 30;10:837741. doi: 10.3389/fped.2022.837741. eCollection 2022. PMID 35433544
- [Derived] Chen L, Tan KML, Gong M, Chong MFF, Tan KH, Chong YS, Meaney MJ, Gluckman PD, Eriksson JG, Karnani N. Variability in newborn telomere length is explained by inheritance and intrauterine environment. BMC Med. 2022 Jan 25;20(1):20. doi: 10.1186/s12916-021-02217-9. PMID 35073935
- [Derived] Wong BW, Toh JY, Sugianto R, Chia A, Tint MT, Yuan WL, Padmapriya N, Lanca C, Saw SM, Lee YS, Shek LP, Tan KH, Yap F, Godfrey KM, Chong YS, Muller-Riemenschneider F, Eriksson JG, Chan SY, Chong MF. Associations of Childcare Arrangements with Adiposity Measures in a Multi-Ethnic Asian Cohort: The GUSTO Study. Int J Environ Res Public Health. 2021 Nov 19;18(22):12178. doi: 10.3390/ijerph182212178. PMID 34831933
- [Derived] Padmapriya N, Chen B, Goh CMJL, Shek LPC, Chong YS, Tan KH, Chan SY, Yap F, Godfrey KM, Lee YS, Eriksson JG, Bernard JY, Muller-Riemenschneider F. 24-hour movement behaviour profiles and their transition in children aged 5.5 and 8 years - findings from a prospective cohort study. Int J Behav Nutr Phys Act. 2021 Nov 6;18(1):145. doi: 10.1186/s12966-021-01210-y. PMID 34742314
- [Derived] Lim IY, Lin X, Teh AL, Wu Y, Chen L, He M, Chan SY, MacIsaac JL, Chan JKY, Tan KH, Chong MFF, Kobor MS, Godfrey KM, Meaney MJ, Lee YS, Eriksson JG, Gluckman PD, Chong YS, Karnani N. Dichotomy in the Impact of Elevated Maternal Glucose Levels on Neonatal Epigenome. J Clin Endocrinol Metab. 2022 Feb 17;107(3):e1277-e1292. doi: 10.1210/clinem/dgab710. PMID 34633450
- [Derived] Ong J, Sadananthan SA, Soh SE, Ng S, Yuan WL, Aris IM, Tint MT, Michael N, Loy SL, Tan KH, Godfrey KM, Shek LP, Yap F, Lee YS, Chong YS, Chan SY. Increasing nausea and vomiting of pregnancy is associated with sex-dependent differences in early childhood growth: the GUSTO mother-offspring cohort study. BMC Pregnancy Childbirth. 2021 Aug 22;21(1):578. doi: 10.1186/s12884-021-04024-9. PMID 34420517
- [Derived] Pang WW, Geddes DT, Lai CT, Chan SY, Chan YH, Cheong CY, Fok D, Chua MC, Lim SB, Huang J, Pundir S, Tan KH, Yap F, Godfrey KM, Gluckman PD, Shek LP, Vickers MH, Eriksson JG, Chong YS, Wlodek ME. The association of maternal gestational hyperglycemia with breastfeeding duration and markers of milk production. Am J Clin Nutr. 2021 Sep 1;114(3):1219-1228. doi: 10.1093/ajcn/nqab142. PMID 33963740
- [Derived] Loo EXL, Lau HX, Suaini NHA, Wong LSY, Goh AEN, Teoh OH, Van Bever HP, Shek LP, Lee BW, Tan KH, Godfrey KM, Eriksson JG, Chong YS, Tham EH. House dust mite sensitization, eczema, and wheeze increase risk of shellfish sensitization. Pediatr Allergy Immunol. 2021 Jul;32(5):1096-1099. doi: 10.1111/pai.13493. Epub 2021 Mar 20. No abstract available. PMID 33687761
- [Derived] van Lee L, Chia A, Phua D, Colega M, Padmapriya N, Bernard JY, Cai S, Tham EKH, Teoh OH, Goh D, Gooley JJ, Gluckman PD, Yap F, Shek LPC, Godfrey KM, Tan KH, Chong YS, Muller-Riemenschneider F, Broekman B, Meaney M, Chen H, Chong MFF. Multiple modifiable lifestyle factors and the risk of perinatal depression during pregnancy: Findings from the GUSTO cohort. Compr Psychiatry. 2020 Nov;103:152210. doi: 10.1016/j.comppsych.2020.152210. Epub 2020 Sep 30. PMID 33045668
- [Derived] Xu J, Lawley B, Wong G, Otal A, Chen L, Ying TJ, Lin X, Pang WW, Yap F, Chong YS, Gluckman PD, Lee YS, Chong MF, Tannock GW, Karnani N. Ethnic diversity in infant gut microbiota is apparent before the introduction of complementary diets. Gut Microbes. 2020 Sep 2;11(5):1362-1373. doi: 10.1080/19490976.2020.1756150. Epub 2020 May 26. PMID 32453615
- [Derived] Tan CW, Sultana R, Kee MZL, Meaney MJ, Sng BL. Investigating the association between labour epidural analgesia and postpartum depression: A prospective cohort study. Eur J Anaesthesiol. 2020 Sep;37(9):796-802. doi: 10.1097/EJA.0000000000001236. PMID 32453169
- [Derived] Tint MT, Sadananthan SA, Soh SE, Aris IM, Michael N, Tan KH, Shek LPC, Yap F, Gluckman PD, Chong YS, Godfrey KM, Velan SS, Chan SY, Eriksson JG, Fortier MV, Zhang C, Lee YS. Maternal glycemia during pregnancy and offspring abdominal adiposity measured by MRI in the neonatal period and preschool years: The Growing Up in Singapore Towards healthy Outcomes (GUSTO) prospective mother-offspring birth cohort study. Am J Clin Nutr. 2020 Jul 1;112(1):39-47. doi: 10.1093/ajcn/nqaa055. PMID 32219421
- [Derived] Fogel A, McCrickerd K, Aris IM, Goh AT, Chong YS, Tan KH, Yap F, Shek LP, Meaney MJ, Broekman BFP, Godfrey KM, Chong MFF, Cai S, Pang WW, Yuan WL, Lee YS, Forde CG. Eating behaviors moderate the associations between risk factors in the first 1000 days and adiposity outcomes at 6 years of age. Am J Clin Nutr. 2020 May 1;111(5):997-1006. doi: 10.1093/ajcn/nqaa052. PMID 32219418
- [Derived] Chen B, Bernard JY, Padmapriya N, Ning Y, Cai S, Lanca C, Tan KH, Yap F, Chong YS, Shek L, Godfrey KM, Saw SM, Chan SY, Eriksson JG, Tan CS, Muller-Riemenschneider F. Associations between early-life screen viewing and 24 hour movement behaviours: findings from a longitudinal birth cohort study. Lancet Child Adolesc Health. 2020 Mar;4(3):201-209. doi: 10.1016/S2352-4642(19)30424-9. Epub 2020 Jan 28. PMID 32004497
- [Derived] Loo EXL, Zhu Y, Lai JS, Chan YH, Ong CN, Tham EH, Goh A, Teoh OH, Tan KH, Yap F, Chong YS, Gluckman PD, Godfrey KM, Van Bever H, Lee BW, Chong MF, Shek LP. Association between maternal carotenoid, vitamin A, and vitamin E levels and allergic outcomes in the offspring in the first 5 years of life. Pediatr Allergy Immunol. 2020 Jan;31(1):95-97. doi: 10.1111/pai.13122. Epub 2019 Oct 9. No abstract available. PMID 31532016
- [Derived] Quah PL, Kleijweg J, Chang YY, Toh JY, Lim HX, Sugianto R, Aris IM, Yuan WL, Tint MT, Bernard JY, Natarajan P, Muller-Riemenschneider F, Godfrey KM, Gluckman PD, Chong YS, Shek LP, Tan KH, Eriksson JG, Yap F, Lee YS, Chong MFF. Association of sugar-sweetened beverage intake at 18 months and 5 years of age with adiposity outcomes at 6 years of age: the Singapore GUSTO mother-offspring cohort. Br J Nutr. 2019 Dec 14;122(11):1303-1312. doi: 10.1017/S0007114519002253. PMID 31477198
- [Derived] Quah PL, Ng JC, Fries LR, Chan MJ, Aris IM, Lee YS, Yap F, Godfrey KM, Chong YS, Shek LP, Tan KH, Forde CG, Chong MFF. Longitudinal Analysis Between Maternal Feeding Practices and Body Mass Index (BMI): A Study in Asian Singaporean Preschoolers. Front Nutr. 2019 Apr 2;6:32. doi: 10.3389/fnut.2019.00032. eCollection 2019. PMID 31001535
- [Derived] Loy SL, Lim LM, Chan SY, Tan PT, Chee YL, Quah PL, Chan JKY, Tan KH, Yap F, Godfrey KM, Shek LP, Chong MF, Kramer MS, Chong YS, Chi C. Iron status and risk factors of iron deficiency among pregnant women in Singapore: a cross-sectional study. BMC Public Health. 2019 Apr 11;19(1):397. doi: 10.1186/s12889-019-6736-y. PMID 30975203
- [Derived] Wu Y, Lin X, Lim IY, Chen L, Teh AL, MacIsaac JL, Tan KH, Kobor MS, Chong YS, Gluckman PD, Karnani N. Analysis of two birth tissues provides new insights into the epigenetic landscape of neonates born preterm. Clin Epigenetics. 2019 Feb 11;11(1):26. doi: 10.1186/s13148-018-0599-4. PMID 30744680
- [Derived] Sadananthan SA, Tint MT, Michael N, Aris IM, Loy SL, Lee KJ, Shek LP, Yap FKP, Tan KH, Godfrey KM, Leow MK, Lee YS, Kramer MS, Gluckman PD, Chong YS, Karnani N, Henry CJ, Fortier MV, Velan SS. Association Between Early Life Weight Gain and Abdominal Fat Partitioning at 4.5 Years is Sex, Ethnicity, and Age Dependent. Obesity (Silver Spring). 2019 Mar;27(3):470-478. doi: 10.1002/oby.22408. Epub 2019 Feb 1. PMID 30707510
- [Derived] Loo EXL, Chew LJM, Zulkifli AB, Ta LDH, Kuo IC, Goh A, Teoh OH, Van Bever H, Gluckman PD, Yap F, Tan KH, Chong YS, Lee BW, Shek LP. Comparison of microbiota and allergen profile in house dust from homes of allergic and non-allergic subjects- results from the GUSTO study. World Allergy Organ J. 2018 Dec 5;11(1):37. doi: 10.1186/s40413-018-0212-5. eCollection 2018. PMID 30534340
- [Derived] Tham EH, Tan PT, Loo EXL, Goh AEN, Teoh OH, Yap F, Tan KH, Godfrey KM, Van Bever HP, Lee BW, Finkelstein EA, Chong YS, Shek LP. Early childcare enrollment and childhood wheezing phenotypes. Pediatr Allergy Immunol. 2019 Feb;30(1):122-127. doi: 10.1111/pai.12983. Epub 2018 Dec 9. No abstract available. PMID 30246437
- [Derived] Bernard JY, Pan H, Aris IM, Moreno-Betancur M, Soh SE, Yap F, Tan KH, Shek LP, Chong YS, Gluckman PD, Calder PC, Godfrey KM, Chong MF, Kramer MS, Karnani N, Lee YS. Long-chain polyunsaturated fatty acids, gestation duration, and birth size: a Mendelian randomization study using fatty acid desaturase variants. Am J Clin Nutr. 2018 Jul 1;108(1):92-100. doi: 10.1093/ajcn/nqy079. PMID 29878044
- [Derived] Soh SE, Goh A, Teoh OH, Godfrey KM, Gluckman PD, Shek LP, Chong YS. Pregnancy Trimester-Specific Exposure to Ambient Air Pollution and Child Respiratory Health Outcomes in the First 2 Years of Life: Effect Modification by Maternal Pre-Pregnancy BMI. Int J Environ Res Public Health. 2018 May 15;15(5):996. doi: 10.3390/ijerph15050996. PMID 29762532
- [Derived] Tham EH, Loo EXL, Goh A, Teoh OH, Yap F, Tan KH, Godfrey KM, Van Bever H, Lee BW, Chong YS, Shek LP. Phototherapy for neonatal hyperbilirubinemia and childhood eczema, rhinitis and wheeze. Pediatr Neonatol. 2019 Feb;60(1):28-34. doi: 10.1016/j.pedneo.2018.03.004. Epub 2018 Mar 24. PMID 29678409
- [Derived] Fogel A, Mccrickerd K, Fries LR, Goh AT, Quah PL, Chan MJ, Toh JY, Chong YS, Tan KH, Yap F, Shek LP, Meaney MJ, Broekman BFP, Lee YS, Godfrey KM, Chong MFF, Forde CG. Eating in the absence of hunger: Stability over time and associations with eating behaviours and body composition in children. Physiol Behav. 2018 Aug 1;192:82-89. doi: 10.1016/j.physbeh.2018.03.033. Epub 2018 Mar 30. PMID 29609000
- [Derived] Chi C, Loy SL, Chan SY, Choong C, Cai S, Soh SE, Tan KH, Yap F, Gluckman PD, Godfrey KM, Shek LP, Chan JKY, Kramer MS, Chong YS. Impact of adopting the 2013 World Health Organization criteria for diagnosis of gestational diabetes in a multi-ethnic Asian cohort: a prospective study. BMC Pregnancy Childbirth. 2018 Mar 21;18(1):69. doi: 10.1186/s12884-018-1707-3. PMID 29562895
- [Derived] Fogel A, Fries LR, McCrickerd K, Goh AT, Quah PL, Chan MJ, Toh JY, Chong YS, Tan KH, Yap F, Shek LP, Meaney MJ, Broekman BFP, Lee YS, Godfrey KM, Fong Chong MF, Forde CG. Oral processing behaviours that promote children's energy intake are associated with parent-reported appetitive traits: Results from the GUSTO cohort. Appetite. 2018 Jul 1;126:8-15. doi: 10.1016/j.appet.2018.03.011. Epub 2018 Mar 15. PMID 29551400
- [Derived] Lim SX, Toh JY, van Lee L, Han WM, Shek LP, Tan KH, Yap F, Godfrey KM, Chong YS, Chong MF. Food Sources of Energy and Macronutrient Intakes among Infants from 6 to 12 Months of Age: The Growing Up in Singapore Towards Healthy Outcomes (GUSTO) Study. Int J Environ Res Public Health. 2018 Mar 10;15(3):488. doi: 10.3390/ijerph15030488. PMID 29534442
- [Derived] Chia AR, Tint MT, Han CY, Chen LW, Colega M, Aris IM, Chua MC, Tan KH, Yap F, Shek LP, Chong YS, Godfrey KM, Fortier MV, Lee YS, Chong MF. Adherence to a healthy eating index for pregnant women is associated with lower neonatal adiposity in a multiethnic Asian cohort: the Growing Up in Singapore Towards healthy Outcomes (GUSTO) Study. Am J Clin Nutr. 2018 Jan 1;107(1):71-79. doi: 10.1093/ajcn/nqx003. PMID 29381790
- [Derived] Lin X, Teh AL, Chen L, Lim IY, Tan PF, MacIsaac JL, Morin AM, Yap F, Tan KH, Saw SM, Lee YS, Holbrook JD, Godfrey KM, Meaney MJ, Kobor MS, Chong YS, Gluckman PD, Karnani N. Choice of surrogate tissue influences neonatal EWAS findings. BMC Med. 2017 Dec 5;15(1):211. doi: 10.1186/s12916-017-0970-x. PMID 29202839
- [Derived] Chen LW, Tint MT, Fortier MV, Aris IM, Shek LP, Tan KH, Chan SY, Gluckman PD, Chong YS, Godfrey KM, Rajadurai VS, Yap F, Kramer MS, Lee YS. Which anthropometric measures best reflect neonatal adiposity? Int J Obes (Lond). 2018 Mar;42(3):501-506. doi: 10.1038/ijo.2017.250. Epub 2017 Oct 9. PMID 28990589
- [Derived] Bernard JY, Padmapriya N, Chen B, Cai S, Tan KH, Yap F, Shek L, Chong YS, Gluckman PD, Godfrey KM, Kramer MS, Saw SM, Muller-Riemenschneider F. Predictors of screen viewing time in young Singaporean children: the GUSTO cohort. Int J Behav Nutr Phys Act. 2017 Sep 5;14(1):112. doi: 10.1186/s12966-017-0562-3. PMID 28870219
- [Derived] Aris IM, Bernard JY, Chen LW, Tint MT, Pang WW, Soh SE, Saw SM, Shek LP, Godfrey KM, Gluckman PD, Chong YS, Yap F, Kramer MS, Lee YS. Modifiable risk factors in the first 1000 days for subsequent risk of childhood overweight in an Asian cohort: significance of parental overweight status. Int J Obes (Lond). 2018 Jan;42(1):44-51. doi: 10.1038/ijo.2017.178. Epub 2017 Jul 28. PMID 28751763
- [Derived] Loy SL, Wee PH, Colega MT, Cheung YB, Aris IM, Chan JKY, Godfrey KM, Gluckman PD, Tan KH, Shek LP, Chong YS, Natarajan P, Muller-Riemenschneider F, Lek N, Rajadurai VS, Tint MT, Lee YS, Chong MF, Yap F. Maternal Night-Fasting Interval during Pregnancy Is Directly Associated with Neonatal Head Circumference and Adiposity in Girls but Not Boys. J Nutr. 2017 Jul;147(7):1384-1391. doi: 10.3945/jn.117.250639. Epub 2017 Jun 7. PMID 28592516
- [Derived] Loo EX, Goh A, Aris IBM, Teoh OH, Shek LP, Lee BW, Chan YH, Tint MT, Soh SE, Saw SM, Gluckman P, Godfrey KM, Chong YS, Yap F, Kramer MS, Van Bever H, Lee YS. Effects of infant weight gain on subsequent allergic outcomes in the first 3 years of life. BMC Pediatr. 2017 Jun 2;17(1):134. doi: 10.1186/s12887-017-0890-0. PMID 28576134
- [Derived] Loo EXL, Sim JZT, Loy SL, Goh A, Chan YH, Tan KH, Yap F, Gluckman PD, Godfrey KM, Van Bever H, Lee BW, Chong YS, Shek LP, Koh MJA, Ang SB. Associations between caesarean delivery and allergic outcomes: Results from the GUSTO study. Ann Allergy Asthma Immunol. 2017 May;118(5):636-638. doi: 10.1016/j.anai.2017.02.021. No abstract available. PMID 28477794
- [Derived] Loy SL, Ng MJH, Cheung YB, Godfrey KM, Calder PC, Lek N, Yap F, Muller-Riemenschneider F, Natarajan P, Chong YS, Tan KH, Shek LP, Chong MF, Chan JKY. Plasma omega-3 fatty acids in pregnancy are inversely associated with postpartum weight retention in a multiethnic Asian cohort. Am J Clin Nutr. 2017 May;105(5):1158-1165. doi: 10.3945/ajcn.116.151258. Epub 2017 Mar 22. PMID 28330907
- [Derived] Pang WW, Colega M, Cai S, Chan YH, Padmapriya N, Chen LW, Soh SE, Han WM, Tan KH, Lee YS, Saw SM, Gluckman PD, Godfrey KM, Chong YS, van Dam RM, Chong MF. Higher Maternal Dietary Protein Intake Is Associated with a Higher Risk of Gestational Diabetes Mellitus in a Multiethnic Asian Cohort. J Nutr. 2017 Apr;147(4):653-660. doi: 10.3945/jn.116.243881. Epub 2017 Mar 8. PMID 28275101
- [Derived] Lin X, Lim IY, Wu Y, Teh AL, Chen L, Aris IM, Soh SE, Tint MT, MacIsaac JL, Morin AM, Yap F, Tan KH, Saw SM, Kobor MS, Meaney MJ, Godfrey KM, Chong YS, Holbrook JD, Lee YS, Gluckman PD, Karnani N; GUSTO study group. Developmental pathways to adiposity begin before birth and are influenced by genotype, prenatal environment and epigenome. BMC Med. 2017 Mar 7;15(1):50. doi: 10.1186/s12916-017-0800-1. PMID 28264723
- [Derived] Fogel A, Goh AT, Fries LR, Sadananthan SA, Velan SS, Michael N, Tint MT, Fortier MV, Chan MJ, Toh JY, Chong YS, Tan KH, Yap F, Shek LP, Meaney MJ, Broekman BFP, Lee YS, Godfrey KM, Chong MFF, Forde CG. A description of an 'obesogenic' eating style that promotes higher energy intake and is associated with greater adiposity in 4.5year-old children: Results from the GUSTO cohort. Physiol Behav. 2017 Jul 1;176:107-116. doi: 10.1016/j.physbeh.2017.02.013. Epub 2017 Feb 14. PMID 28213204
- [Derived] Chen LW, Aris IM, Bernard JY, Tint MT, Colega M, Gluckman PD, Tan KH, Shek LP, Chong YS, Yap F, Godfrey KM, van Dam RM, Chong MF, Lee YS. Associations of maternal macronutrient intake during pregnancy with infant BMI peak characteristics and childhood BMI. Am J Clin Nutr. 2017 Mar;105(3):705-713. doi: 10.3945/ajcn.116.148270. Epub 2017 Feb 8. PMID 28179222
- [Derived] Loy SL, Chan JK, Wee PH, Colega MT, Cheung YB, Godfrey KM, Kwek K, Saw SM, Chong YS, Natarajan P, Muller-Riemenschneider F, Lek N, Chong MF, Yap F. Maternal Circadian Eating Time and Frequency Are Associated with Blood Glucose Concentrations during Pregnancy. J Nutr. 2017 Jan;147(1):70-77. doi: 10.3945/jn.116.239392. Epub 2016 Oct 19. PMID 27798346
- [Derived] Chia AR, de Seymour JV, Colega M, Chen LW, Chan YH, Aris IM, Tint MT, Quah PL, Godfrey KM, Yap F, Saw SM, Baker PN, Chong YS, van Dam RM, Lee YS, Chong MF. A vegetable, fruit, and white rice dietary pattern during pregnancy is associated with a lower risk of preterm birth and larger birth size in a multiethnic Asian cohort: the Growing Up in Singapore Towards healthy Outcomes (GUSTO) cohort study. Am J Clin Nutr. 2016 Nov;104(5):1416-1423. doi: 10.3945/ajcn.116.133892. Epub 2016 Oct 12. PMID 27733407
- [Derived] van Lee L, Tint MT, Aris IM, Quah PL, Fortier MV, Lee YS, Yap FK, Saw SM, Godfrey KM, Gluckman PD, Chong YS, Kramer MS, Chong MF. Prospective associations of maternal betaine status with offspring weight and body composition at birth: the Growing Up in Singapore Towards healthy Outcomes (GUSTO) cohort study. Am J Clin Nutr. 2016 Nov;104(5):1327-1333. doi: 10.3945/ajcn.116.138818. Epub 2016 Sep 21. PMID 27655442
- [Derived] Aris IM, Bernard JY, Chen LW, Tint MT, Pang WW, Lim WY, Soh SE, Saw SM, Godfrey KM, Gluckman PD, Chong YS, Yap F, Kramer MS, Lee YS. Infant body mass index peak and early childhood cardio-metabolic risk markers in a multi-ethnic Asian birth cohort. Int J Epidemiol. 2017 Apr 1;46(2):513-525. doi: 10.1093/ije/dyw232. PMID 27649801
- [Derived] Chen LW, Tint MT, Fortier MV, Aris IM, Bernard JY, Colega M, Gluckman PD, Saw SM, Chong YS, Yap F, Godfrey KM, Kramer MS, van Dam RM, Chong MF, Lee YS. Maternal Macronutrient Intake during Pregnancy Is Associated with Neonatal Abdominal Adiposity: The Growing Up in Singapore Towards healthy Outcomes (GUSTO) Study. J Nutr. 2016 Aug;146(8):1571-9. doi: 10.3945/jn.116.230730. Epub 2016 Jul 6. PMID 27385763
- [Derived] Cheng TS, Loy SL, Toh JY, Cheung YB, Chan JK, Godfrey KM, Gluckman PD, Saw SM, Chong YS, Lee YS, Lek N, Chong MF, Yap F. Predominantly nighttime feeding and weight outcomes in infants. Am J Clin Nutr. 2016 Aug;104(2):380-8. doi: 10.3945/ajcn.116.130765. Epub 2016 Jul 6. PMID 27385614
- [Derived] Quah PL, Cheng TS, Cheung YB, Yap F, Saw SM, Godfrey KM, Gluckman PD, Chong YS, Chong MF. Maternal and infant correlates of maternal feeding beliefs and practices in a multi-ethnic Asian population: the GUSTO (Growing Up in Singapore Towards healthy Outcomes) study. Public Health Nutr. 2016 Oct;19(15):2789-98. doi: 10.1017/S1368980016000744. Epub 2016 Apr 28. PMID 27121890
- [Derived] Tint MT, Fortier MV, Godfrey KM, Shuter B, Kapur J, Rajadurai VS, Agarwal P, Chinnadurai A, Niduvaje K, Chan YH, Aris IB, Soh SE, Yap F, Saw SM, Kramer MS, Gluckman PD, Chong YS, Lee YS. Abdominal adipose tissue compartments vary with ethnicity in Asian neonates: Growing Up in Singapore Toward Healthy Outcomes birth cohort study. Am J Clin Nutr. 2016 May;103(5):1311-7. doi: 10.3945/ajcn.115.108738. Epub 2016 Apr 6. PMID 27053381
- [Derived] Cheng TS, Loy SL, Cheung YB, Chan JK, Pang WW, Godfrey KM, Gluckman PD, Kwek K, Saw SM, Chong YS, Lee YS, Lek N, Yap F. Sexually dimorphic response to feeding mode in the growth of infants. Am J Clin Nutr. 2016 Feb;103(2):398-405. doi: 10.3945/ajcn.115.115493. Epub 2015 Dec 30. PMID 26718413
- [Derived] Quah PL, Chan YH, Aris IM, Pang WW, Toh JY, Tint MT, Broekman BF, Saw SM, Kwek K, Godfrey KM, Gluckman PD, Chong YS, Meaney MJ, Yap FK, van Dam RM, Lee YS, Chong MF; GUSTO Study Group. Prospective associations of appetitive traits at 3 and 12 months of age with body mass index and weight gain in the first 2 years of life. BMC Pediatr. 2015 Oct 12;15:153. doi: 10.1186/s12887-015-0467-8. PMID 26459321
- [Derived] Aris IM, Soh SE, Tint MT, Saw SM, Rajadurai VS, Godfrey KM, Gluckman PD, Yap F, Chong YS, Lee YS. Associations of gestational glycemia and prepregnancy adiposity with offspring growth and adiposity in an Asian population. Am J Clin Nutr. 2015 Nov;102(5):1104-12. doi: 10.3945/ajcn.115.117614. Epub 2015 Sep 30. PMID 26423388
- [Derived] Aris IM, Soh SE, Tint MT, Saw SM, Rajadurai VS, Godfrey KM, Gluckman PD, Yap F, Chong YS, Lee YS. Associations of infant milk feed type on early postnatal growth of offspring exposed and unexposed to gestational diabetes in utero. Eur J Nutr. 2017 Feb;56(1):55-64. doi: 10.1007/s00394-015-1057-0. Epub 2015 Sep 28. PMID 26415764
- [Derived] Chong MF, Ong YL, Calder PC, Colega M, Wong JX, Tan CS, Lim AL, Fisk HL, Cai S, Pang WW, Broekman BF, Saw SM, Kwek K, Godfrey KM, Chong YS, Gluckman P, Meaney MJ, Chen H; GUSTO Study Group. Long-chain polyunsaturated fatty acid status during pregnancy and maternal mental health in pregnancy and the postpartum period: results from the GUSTO study. J Clin Psychiatry. 2015 Jul;76(7):e848-56. doi: 10.4088/JCP.14m09191. PMID 26231011
- [Derived] Lin X, Aris IM, Tint MT, Soh SE, Godfrey KM, Yeo GS, Kwek K, Chan JK, Gluckman PD, Chong YS, Yap F, Holbrook JD, Lee YS. Ethnic Differences in Effects of Maternal Pre-Pregnancy and Pregnancy Adiposity on Offspring Size and Adiposity. J Clin Endocrinol Metab. 2015 Oct;100(10):3641-50. doi: 10.1210/jc.2015-1728. Epub 2015 Jul 22. PMID 26200236
- [Derived] Chong MF, Chia AR, Colega M, Tint MT, Aris IM, Chong YS, Gluckman P, Godfrey KM, Kwek K, Saw SM, Yap F, van Dam RM, Lee YS; GUSTO Study Group. Maternal Protein Intake during Pregnancy Is Not Associated with Offspring Birth Weight in a Multiethnic Asian Population. J Nutr. 2015 Jun;145(6):1303-10. doi: 10.3945/jn.114.205948. Epub 2015 May 6. PMID 25948786
- [Derived] Cai S, Pang WW, Low YL, Sim LW, Sam SC, Bruntraeger MB, Wong EQ, Fok D, Broekman BF, Singh L, Richmond J, Agarwal P, Qiu A, Saw SM, Yap F, Godfrey KM, Gluckman PD, Chong YS, Meaney MJ, Kramer MS, Rifkin-Graboi A; GUSTO Study Group. Infant feeding effects on early neurocognitive development in Asian children. Am J Clin Nutr. 2015 Feb;101(2):326-36. doi: 10.3945/ajcn.114.095414. Epub 2014 Dec 10. PMID 25646330
- [Derived] Aris IM, Gandhi M, Cheung YB, Soh SE, Tint MT, Gluckman PD, Lee YS, Yap FK, Chong YS. A new population-based reference for gestational age-specific size-at-birth of Singapore infants. Ann Acad Med Singap. 2014 Sep;43(9):439-47. PMID 25341628
- [Derived] Chong MF, Wong JX, Colega M, Chen LW, van Dam RM, Tan CS, Lim AL, Cai S, Broekman BF, Lee YS, Saw SM, Kwek K, Godfrey KM, Chong YS, Gluckman P, Meaney MJ, Chen H; GUSTO study group. Relationships of maternal folate and vitamin B12 status during pregnancy with perinatal depression: The GUSTO study. J Psychiatr Res. 2014 Aug;55:110-6. doi: 10.1016/j.jpsychires.2014.04.006. Epub 2014 Apr 16. PMID 24774647
- [Derived] Aris IM, Soh SE, Tint MT, Liang S, Chinnadurai A, Saw SM, Rajadurai VS, Kwek K, Meaney MJ, Godfrey KM, Gluckman PD, Yap FK, Chong YS, Lee YS. Effect of maternal glycemia on neonatal adiposity in a multiethnic Asian birth cohort. J Clin Endocrinol Metab. 2014 Jan;99(1):240-7. doi: 10.1210/jc.2013-2738. Epub 2013 Dec 20. PMID 24243635
- See also: Study website — http://www.gusto.sg